CLINICAL TRIAL: NCT00508183
Title: Single Row Versus Double Row Fixation in Arthroscopic Cuff Repair; a Randomized Controlled Sutdy.
Brief Title: Types of Fixation in Arthroscopic Rotator Cuff Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OHREB2006862-01H
Record Dates: First submitted 2007-07-25; First posted 2007-07-27 (Estimated); Results first posted 2018-01-29 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Rotator Cuff Tear
Keywords: full thickness rotator cuff tear
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single row fixation (Active Comparator)
  Interventions: Procedure: single row
- double row fixation (Active Comparator)
  Interventions: Procedure: double row fixation

INTERVENTIONS:
Procedure: single row — This method involves using a single row of anchor(s) to reattach the cuff to the bone.
  Arms: single row fixation
Procedure: double row fixation — This technique, "double row" fixation, involves adding an extra anchor(s) over the number used for single row fixation. This extra anchor(s) is placed further inside the bone and may help to increase the fixation strength of the repair.
  Arms: double row fixation

SUMMARY:
The study will identify if there is a difference of quality of life after surgery between two techniques used in surgery. The two different techniques are either the Single Row Fixation or the Double Row Fixation.

DETAILED DESCRIPTION:
Primary Research Question; What is the difference in disease specific quality of life between patients who undergo a repair of the rotator cuff with arthroscopic technique using single-row fixation, versus double-row fixation, as measured by the Western Ontario Rotator Cuff Index (WORC)at one year post op?

ELIGIBILITY:
Inclusion Criteria:

* Patients who have failed standard non-surgical management of their rotator cuff tear, and who would benefit from a surgical repair of the cuff.
* Imaging and intra-operative findings confirming a full thickness tear of the rotator cuff.

Exclusion Criteria:

* Characteristics of the cuff tear that render the cuff irrepairable.
* Significant shoulder comorbidities
* Previous surgery on affected shoulder
* Patients with active workers compensation claims
* Active joint or systemic infection
* Significant muscle paralysis
* Rotatorcuff tear arthropathy
* Charcots arthropathy
* Major medical illness
* Unable to speak or read English
* Psychiatric illness that precludes informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lapner, MD, Principal Investigator — OHRI
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

REFERENCES:
- [Result] Lapner PL, Sabri E, Rakhra K, McRae S, Leiter J, Bell K, Macdonald P. A multicenter randomized controlled trial comparing single-row with double-row fixation in arthroscopic rotator cuff repair. J Bone Joint Surg Am. 2012 Jul 18;94(14):1249-57. doi: 10.2106/JBJS.K.00999. PMID 22810395
- [Derived] Lapner P, Li A, Pollock JW, Zhang T, McIlquham K, McRae S, MacDonald P. A Multicenter Randomized Controlled Trial Comparing Single-Row With Double-Row Fixation in Arthroscopic Rotator Cuff Repair: Long-Term Follow-up. Am J Sports Med. 2021 Sep;49(11):3021-3029. doi: 10.1177/03635465211029029. Epub 2021 Aug 16. PMID 34398641

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred from June 2007 to June 2009 at The Ottawa Hospital in Ottawa,Ontario, and the PanAm Clinic in Winnipeg, Manitoba. The target population was men and women of any age with a diagnosis of a full-thickness tear of the rotator cuff according to clinical criteria.
Pre-assignment Details: Nine patients were never randomized because they either postponed or canceled the surgery, and nineteen patients were excluded prior to randomization for other reasons.
Period: Overall Study
Arm/Group | Single Row Fixation | Double Row Fixation
Started | 48 | 42
Completed | 39 | 34
Not Completed | 9 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Row Fixation | Double Row Fixation | Total
Number analyzed (Participants) | 48 | 42 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (8.9) | 57.8 (7) | 56.8 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 35 | 29 | 64
Region of Enrollment [Number; unit: participants] — Ottawa,Ontario Winnipeg, Manitoba
  participants
    Canada | 48 | 42 | 90

OUTCOME MEASURES:

1. Primary Outcome: Western Ontario Rotator Cuff Index (WORC)
Description: Do patients who undergo a repair of the rotator cuff with arthroscopic technique using double row fixation have increased disease specific quality of life (measured by WORC) then patients who undergo a repair with arthroscopic technique using single-row fixation? The WORC scale is from 0% to 100%, with a higher value being indicative of better disease specific quality of life.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Row Fixation | Double Row Fixation
Number analyzed (Participants) | 39 | 34
units on a scale | 84.4 (21.3) | 81.7 (20.9)
Statistical Analysis 1: Comparison: Single Row Fixation vs Double Row Fixation; Test type: Other; p = 0.60, t-test, 2 sided

2. Secondary Outcome: Constant Score
Description: Differences in outcome between the two groups as measured by the Constant score. The constant score ranges from 1 to 100 with a higher value indicative of better shoulder function.
Time Frame: 2 Year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Row Fixation | Double Row Fixation
Number analyzed (Participants) | 39 | 34
units on a scale | 85.6 (14) | 86.3 (14.2)
Statistical Analysis 1: Comparison: Single Row Fixation vs Double Row Fixation; Test type: Other; p = 0.05, t-test, 2 sided

3. Secondary Outcome: ASES Score
Description: Determination of differences in outcome between the two groups as measured by the American Shoulder and Elbow Surgeons (ASES) score. The ASES score ranges from 0 to 100 with a higher number indicative of better function.
Time Frame: 2 Year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Row Fixation | Double Row Fixation
Number analyzed (Participants) | 39 | 34
units on a scale | 87.9 (16.9) | 89.3 (17.5)
Statistical Analysis 1: Comparison: Single Row Fixation vs Double Row Fixation; Test type: Other; p = 0.05, t-test, 2 sided

4. Secondary Outcome: Strength Test
Description: Shoulder strength in forward elevation was measured in kg using a portable scale.
Time Frame: 2 Years
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Single Row Fixation | Double Row Fixation
Number analyzed (Participants) | 39 | 34
kg | 8.0 (6) | 7.3 (3.2)

5. Secondary Outcome: Healing Rate
Description: Percentage of Participants who had healed by 1 year post-surgery as measured using magnetic resonance imaging. If the tendons were in continuity with no evidence of full-thickness tearing, the repair was considered healed (intact).
Time Frame: 1 Year
Measure: Number; unit: percentage of patients
Arm/Group | Single Row Fixation | Double Row Fixation
Number analyzed (Participants) | 39 | 34
percentage of patients | 67 | 78
Statistical Analysis 1: Comparison: Single Row Fixation vs Double Row Fixation; Test type: Other; p = 0.05, Chi-squared

ADVERSE EVENTS:
Arm/Group | Single Row Fixation | Double Row Fixation
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/42
Other Adverse Events (participants affected / at risk) | 0/48 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No